CLINICAL TRIAL: NCT02549703
Title: Mitochondrial Dysfunction and Disease Progression
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Columbia University (Other); New York Stem Cell Foundation Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1495; CDMRP-MS140072 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Clinically Isolated Syndrome; Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
Keywords: multiple sclerosis; progressive multiple sclerosis; mitochondria; neurodegeneration
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and CSF samples will be stored indefinitely at the Casaccia lab. Skin samples will be stored indefinitely at the New York Stem Cell Foundation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Relapsing Remitting Multiple Sclerosis: Patients with Relapsing Remitting Multiple Sclerosis/Clinically Isolated Syndrome
- Secondary Progressive Multiple Sclerosis
- Primary Progressive Multiple Sclerosis

SUMMARY:
While the last several years have seen great strides in the treatment of relapsing forms of MS, progressive MS, responsible for the majority of MS-related disability, lags far behind. Despite much research, the lack of understanding related to what causes patients' relentless decline in function results in an inability to develop targeted treatment strategies suitable for clinical trials. This grant has two main goals.

The first goal is to extend the investigators preliminary study on rat neurons treated with the CSF of MS patients to a larger number of Progressive patients in order to validate the initial findings and extend the study to include analysis of human neurons. The initiating PI (Dr. Casaccia) and the Partnering PI and Clinical Neurologist (Dr. Katz Sand) have recently identified components that are present in the CSF of progressive patients that impair the ability of rat neurons to produce energy. The partnering PI, Dr. Quinzii (Columbia University) together with collaborator Dr. Fossati (NY Stem Cells Foundation), have characterized human neurons generated from stem cells derived from skin biopsies of progressive patients and detected the presence of energetic deficits. The experimental plan will build on these results and test hypotheses of disease progression. The overall goal is to improve understanding on how to stop neurons from degenerating and stop clinical progression.

The second goal is to ask whether it is possible to define a progressive disease course on the basis of combined biochemical, functional and imaging measurements. The initiating PI will be responsible for the biochemical assessment of CSF and serum samples and, together with partnering PI Quinzii, will also provide functional bioassays measurements of mitochondrial bioenergetics impairment in patients. These data will be combined with clinical assessment and MRI evaluations conducted by the partnering PI Katz Sand and collaborator Inglese. A two year clinical and imaging follow up from the initial recruitment will allow to define whether the combined measurements can be used by clinical neurologists to define the disease course and better identify therapeutic options for patients.

The expectation is that the completion of the stated aims of research will allow an advancement of the current knowledge of the progressive form of MS and lead to potential new therapeutic targets.

ELIGIBILITY:
Inclusion criteria:

* male and female subjects age 18 or older
* diagnosis of one of the following:

  1. RRMS according to McDonald 2010 criteria or a diagnosis of CIS with clinical symptoms and MRI consistent with MS
  2. PPMS according to McDonald 2010 criteria
  3. SPMS defined as at least six months of progressive decline following an initial relapsing disease course
* able and willing to undergo clinical evaluation, MRI, lumbar puncture, and skin biopsy and to return for follow up assessments at the end of year 1 and year 2
* able and willing to provide informed consent.

Exclusion criteria:

* pregnancy
* inability to undergo lumbar puncture, due to anticoagulant therapy that cannot be held for the day of the procedure or results of screening laboratory testing or the presence of another medical condition that would render the procedure unsafe, as determined by the investigator
* inability to undergo MRI, due to the presence of metallic implants incompatible with MRI or any other reason
* presence of other severe medical conditions likely to influence study results or that raise the likelihood of harm to the patient as a result of study participation, as determined by the investigator (e.g. the presence of a brain mass, which could influence the CSF results and also might make lumbar puncture unsafe)
* inability to complete the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients willing and able to undergo the assessments required for this study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Spare respiratory capacity | 2 years
  Mitochondrial bioenergetic measurements
Oxygen consumption rate | 2 years
  Mitochondrial bioenergetic measurements

SECONDARY OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC) Score | 1 year
  MS disease progression as measured by MSFC score which consists of the Timed 25-foot walk (T25FW) as a measure of ambulation, the Nine-hole peg test (9HPT) as a measure of arm and hand function.
Multiple Sclerosis Functional Composite (MSFC) Score | 2 years
  MS disease progression as measured by MSFC score which consists of the Timed 25-foot walk (T25FW) as a measure of ambulation, the Nine-hole peg test (9HPT) as a measure of arm and hand function.
Expanded Disability Status Scale | 2 years
  a formalized version of the neurological examination
MS Impact Scale-29 (MSIS-29) | 2 years
  a quality of life measure; an overall measure of functioning from the patient's perspective

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Katz Sand, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine, New York, New York, United States